CLINICAL TRIAL: NCT03899259
Title: A Multicenter, Randomized, Double-Blind, Placebo- Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients With Severe or Very Severe Alopecia Areata
Brief Title: A Study of Baricitinib (LY3009104) in Adults With Severe or Very Severe Alopecia Areata
Acronym: BRAVE-AA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16978; I4V-MC-JAIR (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 4 Milligram (mg) Baricitinib (Experimental): Participants received one 4 mg Baricitinib tablet administered orally, every day (QD) one placebo tablet administered orally QD to maintain blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 2 mg Baricitinib (Experimental): Participants received one 2 mg Baricitinib tablet administered orally QD, and one placebo tablet administered orally QD to maintain blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo (Placebo Comparator): Participants received two placebo tablets administered orally QD to maintain the blind.
  Interventions: Drug: Placebo
- 4 mg Baricitinib Maximum Extended Enrollment (MEE) (Experimental): Participants received one 4 mg Baricitinib tablet administered orally, every day (QD) one placebo tablet administered orally QD to maintain blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 2 mg Baricitinib MEE (Experimental): Participants received one 2 mg Baricitinib tablet administered orally QD, and one placebo tablet administered orally QD to maintain blind.
  Interventions: Drug: Baricitinib
- Placebo MEE (Placebo Comparator): Participants received two placebo tablets administered orally QD to maintain the blind.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: 2 mg Baricitinib; 2 mg Baricitinib MEE; 4 Milligram (mg) Baricitinib; 4 mg Baricitinib Maximum Extended Enrollment (MEE)
Drug: Placebo — Administered orally
  Arms: 2 mg Baricitinib; 4 Milligram (mg) Baricitinib; 4 mg Baricitinib Maximum Extended Enrollment (MEE); Placebo; Placebo MEE

SUMMARY:
The reason for this study is to see if baricitinib is safe and effective in adults with severe or very severe alopecia areata (AA).

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years and ≤60 years for males (≤70 years of age for females) at the time of informed consent.
* Have severe or very severe AA, as determined by all of the following:

  * Current AA episode of more than 6 months' duration and hair loss encompassing ≥50% of the scalp, as measured by SALT (AA-IGA of 3 or 4) at screening and baseline.
  * No spontaneous improvement over the past 6 months.
  * Current episode of severe or very severe AA of less than 8 years. Note: participants who have severe or very severe AA for ≥8 years may be enrolled if episodes of regrowth, spontaneous or under treatment, have been observed on the affected areas over the past 8 years.
* Male or nonpregnant, nonbreastfeeding female participants.

Exclusion Criteria:

* Primarily "diffuse" type of AA.
* Are currently experiencing other forms of alopecia or any other concomitant conditions that would interfere with evaluations of the effect of study medication on AA.
* Previously treated with an oral Janus kinase (JAK) inhibitor and had an inadequate response (for example, absence of significant terminal hair growth after at least 12 weeks of treatment).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2024-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM -5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (96):
- United States (33):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Investigate MD, Scottsdale, Arizona
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Quest Dermatology Research, Northridge, California
  - Kaiser Permanente Hospital, San Francisco, California
  - New England Research Associates, Bridgeport, Connecticut
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - New Horizon Research Center, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Dermatology and Skin Cancer Specialists, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Associated Skin Care Specialists, New Brighton, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Joseph J. Schwartz, M.D., Troy, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Dermatology Specialists of Charlotte, Charlotte, North Carolina
  - M3-Emerging Medical Research, Raleigh, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Dermatologists of Southwest Ohio, Mason, Ohio
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Northwest Dermatology Institute, Portland, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Argentina (7):
  - Stat Research, CABA, Buenos Aires
  - Instituto de Neumonología y Dermatología, Capital Federal, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Buenos Aires Skin, Buenos Aires, Buenos Aires F.D.
  - Fundacion Respirar, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - Parra Dermatología, Mendoza
- Australia (7):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Skin & Cancer Foundation Australia, Westmead, New South Wales
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Clinical Trials SA Pty Ltd, Campbelltown, South Australia
  - Skin Health Institute Inc., Carlton, Victoria
  - Sinclair Dermatology, Melbourne, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Brazil (8):
  - IDERJ - Instituto de Dermatologia e Estética do Brasil, Rio de Janeiro, Rio de Janeiro
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Hospital de Clínicas Da Universidade Estadual de Campinas, Campinas, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - IPITEC, São Paulo
  - Servidor Público Estadual - IAMSPE - centro de estudos urológicos, São Paulo
- China (15):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Guangdong Province Dermatology Hospital, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - HuaShan Hospital Affiliated To Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Israel (7):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Emek Medical Center, Afula, Northern District
  - Rambam Medical Center, Haifa, Northern District
  - Soroka Medical Center, Beersheba, Southern District
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
- Japan (8):
  - Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Koto-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Tokyo Medical Univ. Hospital, Shinjuku-ku, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Osaka City University Hospital, Osaka
- Clinical Research Puerto Rico, San Juan, Puerto Rico
- South Korea (6):
  - Dankook University Hospital, Cheonan, Chungcheongnam-do
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Boramae Medical Center, Dongjak-gu, Seoul-teukbyeolsi [Seoul]
  - Kyunghee University Hospital at Gangdong, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (4):
  - Chung Shan Medical University Hospital, Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] King B, Mostaghimi A, Shimomura Y, Piraccini BM, Blume-Peytavi U, Sontag A, Dutronc Y, Denning K, Kolodsick J, Lu X, Srivastava A, Sinclair R. Safety of Baricitinib in Adults with Severe Alopecia Areata from Two Phase III Trials Over a Median of 2.3 Years and Up to 4 Years of Treatment. Am J Clin Dermatol. 2025 Jul;26(4):611-622. doi: 10.1007/s40257-025-00932-0. Epub 2025 Apr 11. PMID 40214720
- [Derived] Craiglow B, Lee YW, Vano-Galvan S, Egeberg A, Dutronc Y, Durand F, Pierce E, Yu G, Chen YF, Mostaghimi A. Improvement in Measures of Quality of Life and Symptoms of Anxiety and Depression in Patients with Severe Alopecia Areata Achieving Sustained Scalp Hair Regrowth with Baricitinib. Dermatol Ther (Heidelb). 2024 Jul;14(7):1959-1968. doi: 10.1007/s13555-024-01208-x. Epub 2024 Jun 21. PMID 38904749
- [Derived] Senna MM, Kwon O, Piraccini BM, Sinclair R, Ball S, Ding Y, Chen YF, Dutronc Y, King B. Clinical Benefits of Baricitinib Therapy According to Scalp Hair Regrowth in Patients with Severe Alopecia Areata. Dermatol Ther (Heidelb). 2023 Dec;13(12):3209-3220. doi: 10.1007/s13555-023-01063-2. Epub 2023 Nov 22. PMID 37991697
- [Derived] Ko JM, Mayo TT, Bergfeld WF, Dutronc Y, Yu G, Ball SG, Somani N, Craiglow BG. Clinical Outcomes for Uptitration of Baricitinib Therapy in Patients With Severe Alopecia Areata: A Pooled Analysis of the BRAVE-AA1 and BRAVE-AA2 Trials. JAMA Dermatol. 2023 Sep 1;159(9):970-976. doi: 10.1001/jamadermatol.2023.2581. PMID 37556146
- [Derived] Piraccini BM, Ohyama M, Craiglow B, Bewley A, Ding Y, Chen YF, Dutronc Y, Pierce E, Durand F, Mostaghimi A. Scalp hair regrowth is associated with improvements in health-related quality of life and psychological symptoms in patients with severe alopecia areata: results from two randomized controlled trials. J Dermatolog Treat. 2023 Dec;34(1):2227299. doi: 10.1080/09546634.2023.2227299. PMID 37381691
- [Derived] Kwon O, Senna MM, Sinclair R, Ito T, Dutronc Y, Lin CY, Yu G, Chiasserini C, McCollam J, Wu WS, King B. Efficacy and Safety of Baricitinib in Patients with Severe Alopecia Areata over 52 Weeks of Continuous Therapy in Two Phase III Trials (BRAVE-AA1 and BRAVE-AA2). Am J Clin Dermatol. 2023 May;24(3):443-451. doi: 10.1007/s40257-023-00764-w. Epub 2023 Mar 1. PMID 36855020
- [Derived] King B, Mostaghimi A, Shimomura Y, Zlotogorski A, Choi GS, Blume-Peytavi U, Passeron T, Holzwarth K, Dutronc Y, McCollam J, Yang FE, Stanley S, Wu WS, Sinclair R. Integrated safety analysis of baricitinib in adults with severe alopecia areata from two randomized clinical trials. Br J Dermatol. 2023 Feb 10;188(2):218-227. doi: 10.1093/bjd/ljac059. PMID 36763878
- [Derived] King B, Ohyama M, Kwon O, Zlotogorski A, Ko J, Mesinkovska NA, Hordinsky M, Dutronc Y, Wu WS, McCollam J, Chiasserini C, Yu G, Stanley S, Holzwarth K, DeLozier AM, Sinclair R; BRAVE-AA Investigators. Two Phase 3 Trials of Baricitinib for Alopecia Areata. N Engl J Med. 2022 May 5;386(18):1687-1699. doi: 10.1056/NEJMoa2110343. Epub 2022 Mar 26. PMID 35334197
- See also: A Study of Baricitinib (LY3009104) in Adults With Severe or Very Severe Alopecia Areata — https://trials.lillytrialguide.com/en-US/trial/10fuouLYVPNjWekNxnfJoE

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results for maximum extended enrollment (MEE) participants will be posted after the study completion.
Groups:
- 4 mg Baricitinib: Participants received one 4 mg Baricitinib administered orally every day (QD) and one placebo administered orally QD to maintain blind.
Period: Overall Study
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Started | 156 | 156 | 234
Received at Least One Dose of Study Drug | 155 | 156 | 234
Completed | 0 | 0 | 0
Not Completed | 156 | 156 | 234
Not completed — Adverse Event | 5 | 4 | 6
Not completed — Lack of Efficacy | 5 | 0 | 2
Not completed — Pregnancy | 3 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Deviation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 8 | 10 | 12
Not completed — Lost to Follow-up | 5 | 6 | 2
Not completed — Lack of Adherence | 1 | 0 | 0
Not completed — Screen Failure | 1 | 0 | 0
Not completed — Ongoing Study Participation | 127 | 134 | 210

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib | Total
Number analyzed (Participants) | 156 | 156 | 234 | 546
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant was randomized inadvertently but not dosed and age was not obtained.
  years
    number analyzed (Participants) | 155 | 156 | 234 | 545
    (all) | 37.10 (12.35) | 39.00 (12.99) | 38.00 (12.65) | 38.00 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 103 | 144 | 345
  Male | 58 | 53 | 90 | 201
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 51 | 49 | 67 | 167
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 16 | 12 | 18 | 46
  White | 85 | 92 | 144 | 321
  More than one race | 4 | 2 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 15 | 11 | 20 | 46
  Australia | 17 | 17 | 20 | 54
  Brazil | 14 | 13 | 24 | 51
  China | 2 | 2 | 6 | 10
  Israel | 14 | 19 | 25 | 58
  Japan | 10 | 11 | 20 | 41
  South Korea | 23 | 17 | 26 | 66
  Taiwan | 7 | 12 | 11 | 30
  United States | 54 | 54 | 82 | 190
Baseline Disease Severity of Alopecia Tool (SALT) Score [Mean (Standard Deviation); unit: units on a scale] — SALT uses a visual aid showing the division of the scalp hair into 4 areas - top of the head constituting 40% of total surface, the posterior/back of head 24%, right and left side of head 18% each. The percentage of hair loss in each area is determined and is multiplied by the percentage of scalp covered by that area. The total sum of the 4 products of each area will give the SALT score. Only terminal hair is included in the SALT; vellus hair or any fine downy hair is not taken into account for scoring. The score will range from 0% to 100%, with lower score indicating better health outcomes.
  units on a scale | 85 (17.79) | 85.6 (18.08) | 84.8 (18.08) | 85.1 (17.97)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Severity of Alopecia Tool (SALT) ≤ 20
Description: The SALT uses a visual aid showing the division of the scalp hair into 4 areas with the top of the head constituting 40% of total surface, the posterior/back of head 24%, right side and left side of head 18% each. The percentage of hair loss in each area is determined and is multiplied by the percentage of scalp covered by that area. The total sum of the 4 products of each area will give the SALT score, as developed by the National Alopecia Areata Foundation Working Committee. Only terminal hair is included in the SALT; vellus hair or any fine downy hair is not taken into account in the SALT scoring process. The SALT score will range from 0% to 100%, with lower score indicating better health outcomes.
Time Frame: Week 36
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 156 | 156 | 234
percentage of participants | 2.6 [1.0 to 6.4] | 17.3 [12.2 to 24.0] | 32.5 [26.8 to 38.7]
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.86, 95% CI 2-sided [2.79 to 22.17]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 19.72, 95% CI 2-sided [7.30 to 53.30]

2. Secondary Outcome: Percent Change From Baseline in SALT Score at Week 36
Description: SALT uses a visual aid showing the division of the scalp hair into4 areas with the top of the head constituting 40% of total surface, the posterior/back of head 24%, right side and left side of head 18% each. The percentage of hair loss in each area is determined and is multiplied by the percentage of scalp covered by that area. The total sum of the 4 products of each area will give the SALT score. Only terminal hair is included in the SALT; vellus hair or any fine downy hair is not taken into account in the SALT scoring process. The SALT score will range from 0% to 100%, with lower score indicating better health outcomes. Least Squares Mean (LSM) was calculated using analysis of covariance (ANCOVA) with geographic region duration of current episode at baseline (< 4 years versus ≥4 years), treatment group, and baseline value in the model.
Time Frame: Baseline, Week 36
Population: All randomized participants with nonmissing baseline and at least one postbaseline measure. The method used to handle missing data was modified last observation carried forward (mLOCF) which used the most recent nonmissing postbaseline assessment.
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Groups:
- 4 mg Baricitinib: Participants received one 4 mg Baricitinib tablet administered orally, every day (QD) one placebo tablet administered orally QD to maintain blind.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 153 | 151 | 230
percentage of change | -2.96 (2.723) | -28.21 (2.770) | -47.45 (2.229)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -25.25, 95% CI 2-sided [-32.78 to -17.72], Standard Error of Mean 3.834
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -44.49, 95% CI 2-sided [-51.33 to -37.65], Standard Error of Mean 3.482

3. Secondary Outcome: Percentage of Participants Achieving 50% Improvement of Severity of Alopecia Tool (SALT50)
Description: SALT uses a visual aid showing the division of the scalp hair into 4 areas with the top of the head constituting 40% of total surface, the posterior/back of head 24%, right side and left side of head 18% each. The percentage of hair loss in each area is determined and is multiplied by the percentage of scalp covered by that area. The total sum of the 4 products of each area will give the SALT score, as developed by the National Alopecia Areata Foundation Working Committee. Only terminal hair is included in the SALT; vellus hair or any fine downy hair is not taken into account in the SALT scoring process. The SALT score will range from 0% to 100%, with lower score indicating better health outcomes. SALT50 indicates at least a 50 % improvement from baseline in the SALT score.
Time Frame: Week 12
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 156 | 156 | 234
percentage of participants | 2.6 [1.0 to 6.4] | 10.9 [6.9 to 16.8] | 23.5 [18.5 to 29.3]
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 4.63, 95% CI 2-sided [1.58 to 13.60]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 12.94, 95% CI 2-sided [4.72 to 35.44]

4. Secondary Outcome: Percentage of Participants With Patient-Reported Outcome (PRO) for Scalp Hair Assessment Score of 0 or 1 With a ≥2-point Improvement From Baseline Among Participants With a Score of ≥3 at Baseline
Description: PRO is an assessment of the particpant's current extent of scalp involvement. It is comprised of 5 category response options: 0= No missing hair (0% of my scalp is missing hair; I have a full head of hair); 1 = A limited area (1% to 20% of my scalp is missing hair); 2 = A moderate area (21% to 49% of my scalp is missing hair); 3 = A large area (50% to 94% of my scalp is missing hair); and 4 = Nearly all or all (95% to 100% of my scalp is missing hair).
Time Frame: Week 36
Population: All randomized participants with baseline PRO for scalp hair assessment score of ≥ 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 4 mg Baricitinib: Participants received one 4 mg Baricitinib tablet administered orally QD, one placebo tablet administered orally QD to maintain blind.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 151 | 149 | 215
percentage of participants | 4.0 [1.8 to 8.4] | 16.1 [11.1 to 22.8] | 34.4 [28.4 to 41.0]
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 4.36, 95% CI 2-sided [1.77 to 10.74]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 13.37, 95% CI 2-sided [5.75 to 31.10]

5. Secondary Outcome: Time for Participants to Achieve SALT ≤ 20
Description: Time for participants to achieve SALT ≤ 20
Time Frame: Week 52
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Percentage of Participants Achieving Clinician-Reported Outcome (ClinRO) Measure for Eyebrow (EB) Hair Loss 0 or 1 With ≥2-point Improvement From Baseline (Among Participants With ClinRO Measure for EB Hair Loss ≥2 at Baseline)
Description: ClinRO is a clinician reported assessment which measures a participant's EB hair loss. It is comprised of 4 category response options: 0 = EB have full coverage and no areas of hair loss; 1 = There are minimal gaps in EB hair and distribution is even; 2 = There are significant gaps in EB hair or distribution is not even; 3 = No notable EB.
Time Frame: Week 36
Population: All randomized participants with baseline ClinRO measure for EB hair loss ≥ 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 112 | 104 | 161
percentage of participants | 4.5 [1.9 to 10.0] | 11.5 [6.7 to 19.1] | 34.8 [27.9 to 42.4]
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.076, Regression, Logistic; Odds Ratio (OR) = 2.56, 95% CI 2-sided [0.91 to 7.24]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.30, 95% CI 2-sided [4.12 to 25.77]

7. Secondary Outcome: Percentage of Participants Achieving ClinRO Measure for Eyelash (EL) Hair Loss 0 or 1 With ≥2-point Improvement From Baseline (Among Participants With ClinRO Measure for EL Hair Loss ≥2 at Baseline)
Description: ClinRO measure for EL hair loss is comprised of 4 category response options: 0 = The EL form a continuous line along the eyelids on both eyes; 1 = There are minimal gaps and the EL are evenly spaced along the eyelids on both eyes; 2 = There are significant gaps along the eyelids or the EL are not evenly spaced along the eyelids; 3 = No notable EL.
Time Frame: Week 36
Population: All randomized participants with baseline ClinRO measure for EL hair loss ≥ 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 90 | 89 | 140
percentage of participants | 5.6 [2.4 to 12.4] | 10.1 [5.4 to 18.1] | 34.3 [26.9 to 42.5]
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.260, Regression, Logistic; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.63 to 5.62]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.10, 95% CI 2-sided [3.18 to 20.66]

8. Secondary Outcome: Percentage of Participants Achieving Patient-Reported Outcome (PRO) Measure for EB 0 or 1 With ≥2-point Improvement From Baseline (Among Participants With PRO Measure for EB ≥2 at Baseline)
Description: PRO is an assessment of the participant's current appearance of eyebrows. It is comprised of 4 category response options: 0 = I have full EB on each eye; 1= I have a minimal gap(s) or a minimal amount of thinning in at least 1 of my EB; 2 = I have a large gap(s) or a large amount of thinning in at least 1 of my EB; and 3 = I have no or barely any EB hairs.
Time Frame: Week 36
Population: All randomized participants with baseline PRO measures for EB hair loss ≥2.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 107 | 108 | 165
percentage of participants | 4.7 [2.0 to 10.5] | 14.8 [9.3 to 22.7] | 35.8 [28.8 to 43.3]
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.017, Regression, Logistic; Odds Ratio (OR) = 3.43, 95% CI 2-sided [1.25 to 9.40]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.85, 95% CI 2-sided [4.32 to 27.25]

9. Secondary Outcome: Percentage of Participants Achieving PRO Measure for EL 0 or 1 With ≥2-point Improvement From Baseline (Among Participants With PRO Measure EL ≥2 at Baseline)
Description: PRO assessment of the participant's current appearance of EL. It is comprised of 4 category response options: 0 = I have full EL on each eyelid; 1 = I have a minimal gap or minimal gaps along the eyelids; 2 = I have a large gap or large gaps along the eyelids; and 3 = I have no or barely any EL hair.
Time Frame: Week 36
Population: All randomized participants with baseline PRO Measure EL hair loss ≥2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 89 | 90 | 133
percentage of participants | 1.1 [0.2 to 6.1] | 18.9 [12.1 to 28.2] | 34.6 [27.0 to 43.0]
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 14.63, 95% CI 2-sided [2.73 to 78.42]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 30.37, 95% CI 2-sided [5.93 to 99.99]

10. Secondary Outcome: Change From Baseline in Skindex-16 Alopecia Areata (AA) Symptoms Domain Score
Description: Skindex-16 AA was adapted from Skindex-16 for use among adults with alopecia areata. It examines the degree to which the participant is bothered by alopecia (hair loss) and associated symptoms. It is composed of 16 items grouped under 3 domains: Symptoms (4 items), Emotions (7 items), and Functioning (5 items). The score of each item ranges from 0 (never bothered) to 6 (always bothered). Symptoms domain score is sum of 4 items, range 0 to 24; Emotions domain score is sum of 7 items, range 0 to 42; Functioning score is sum of 5 items, range 0 to 30. Higher scores indicate a greater impact on quality of life.
  LS means was calculated using the ANCOVA model with geographic region, duration of current episode at Baseline (<4 years vs. ≥ 4years), treatment group, and baseline value as fixed factors.
Time Frame: Baseline, Week 36
Population: All randomized participants with baseline and at least one postbaseline Skindex-16 AA Symptoms Domain Score. The method used to handle missing data was modified last observation carried forward (mLOCF) which used the most recent nonmissing postbaseline assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 146 | 147 | 227
score on a scale | 1.17 (1.415) | -1.85 (1.425) | -3.04 (1.138)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.129, ANCOVA; Mean Difference (Final Values) = -3.02, 95% CI 2-sided [-6.91 to 0.88], Standard Error of Mean 1.981
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.020, ANCOVA; Mean Difference (Final Values) = -4.21, 95% CI 2-sided [-7.75 to -0.68], Standard Error of Mean 1.799

11. Secondary Outcome: Change From Baseline in Skindex-16 AA Emotions Domain Score at Week 36
Description: as for outcome 10
Time Frame: Baseline, Week 36
Population: All randomized participants with baseline and at least one postbaseline Skindex-16 AA emotions domain score. The method used to handle missing data was modified last observation carried forward (mLOCF) which used the most recent nonmissing postbaseline assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- 4 mg Baricitinib: Participants received one 4 mg Baricitinib tablet administered orally, QD one placebo tablet administered orally QD to maintain blind.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 146 | 147 | 227
score on a scale | -11.98 (2.154) | -18.73 (2.171) | -25.40 (1.732)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.026, ANCOVA; Mean Difference (Final Values) = -6.75, 95% CI 2-sided [-12.68 to -0.82], Standard Error of Mean 3.017
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -13.42, 95% CI 2-sided [-18.80 to -8.04], Standard Error of Mean 2.737

12. Secondary Outcome: Change From Baseline in Skindex-16 AA Functioning Domain Score at Week 36
Description: as for outcome 10
Time Frame: Baseline, Week 36
Population: All randomized participants with baseline and at least one postbaseline Skindex-16 AA functioning domain score. The method used to handle missing data was modified last observation carried forward (mLOCF) which used the most recent nonmissing postbaseline assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- 4 mg Baricitinib: Participants received one 4 mg Baricitinib tablet administered orally QD, and one placebo tablet administered orally QD to maintain blind.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 146 | 147 | 227
score on a scale | -9.67 (1.913) | -14.05 (1.925) | -18.00 (1.535)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.103, ANCOVA; Mean Difference (Final Values) = -4.38, 95% CI 2-sided [-9.65 to 0.88], Standard Error of Mean 2.680
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -8.33, 95% CI 2-sided [-13.10 to -3.56], Standard Error of Mean 2.429

13. Secondary Outcome: Mean Change From Baseline in Hospital Anxiety Depression Scale (HADS) Anxiety Score at Week 36
Description: The HADS is a 14-item self-assessment scale that determines the levels of anxiety and depression that a patient is experiencing over the past week. The HADS utilizes a 4-point Likert scale (for example, 0 to 3) for each question and is intended for ages 12 to 65 years. Scores for each domain (anxiety and depression) can range from 0 to 21, with higher scores indicating greater anxiety or depression.
  LS mean was calculated using an ANCOVA model which includes geographic region, duration of current episode at baseline (<4 years vs. ≥4 years), treatment group and baseline score as fixed factors.
Time Frame: Baseline, Week 36
Population: All randomized participants with baseline and at least one postbaseline HADS anxiety score. The method used to handle missing data was modified last observation carried forward (mLOCF) which used the most recent nonmissing postbaseline assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 146 | 147 | 227
score on a scale | -0.47 (0.225) | -0.67 (0.227) | -1.19 (0.181)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.518, ANCOVA; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.82 to 0.42], Standard Error of Mean 0.315
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.012, ANCOVA; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.28 to -0.16], Standard Error of Mean 0.286

14. Secondary Outcome: Mean Change From Baseline in HADS Depression Score at Week 36
Description: as for outcome 13
Time Frame: Baseline,Week 36
Population: All randomized participants with baseline and at least one postbaseline HADS depression score. The method used to handle missing data was modified last observation carried forward (mLOCF) which used the most recent nonmissing postbaseline assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 144 | 156 | 234
score on a scale | 0.29 (0.208) | -0.22 (0.210) | -0.39 (0.167)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.083, ANCOVA; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.08 to 0.07], Standard Error of Mean 0.291
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.010, ANCOVA; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.20 to -0.16], Standard Error of Mean 0.264

ADVERSE EVENTS:
Time Frame: Baseline Up to 36 Weeks
Description: All randomized participants who received at least one dose of study drug, and did not discontinue from the study for the reason "Lost to Follow-up" at the first postbaseline visit.
  Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/155 | 0/233
Serious Adverse Events (participants affected / at risk) | 3/154 | 4/155 | 8/233
Other Adverse Events (participants affected / at risk) | 28/154 | 39/155 | 63/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=154) | 2 mg Baricitinib (N=155) | 4 mg Baricitinib (N=233)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sars-cov-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/57 (1) | 0/53 (0) | 0/89 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=154) | 2 mg Baricitinib (N=155) | 4 mg Baricitinib (N=233)
Nasopharyngitis (Infections and infestations) | 7 (7) | 2 (3) | 15 (19)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 12 (13) | 15 (16)
Urinary tract infection (Infections and infestations) | 2 (2) | 12 (14) | 11 (14)
Headache (Nervous system disorders) | 10 (11) | 12 (15) | 21 (28)
Acne (Skin and subcutaneous tissue disorders) | 3 (4) | 9 (10) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT03899259/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT03899259/SAP_001.pdf